CLINICAL TRIAL: NCT03772587
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of M281 Administered to Adults With Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of M281 Administered to Adults With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOM-M281-004; 2018-002247-28 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Generalized Myasthenia Gravis
Keywords: M281; Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Placebo Comparator)
  Interventions: Other: Placebo
- Group 2 (Experimental)
  Interventions: Drug: M281
- Group 3 (Experimental)
  Interventions: Drug: M281
- Group 4 (Experimental)
  Interventions: Drug: M281
- Group 5 (Experimental)
  Interventions: Drug: M281

INTERVENTIONS:
Drug: M281 — M281 administered as IV infusion
  Arms: Group 2; Group 3; Group 4; Group 5
Other: Placebo — Placebo administered as intravenous (IV) infusion
  Arms: Group 1

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of M281 administered to participants with generalized myasthenia gravis (gMG) who have an insufficient clinical response to ongoing standard of care therapy.

ELIGIBILITY:
Participants must be ≥18 years of age with a documented history of Generalized Myasthenia Gravis (gMG) and clinical signs/symptoms of gMG, not pregnant or breastfeeding, and no history of any neurologic disorder other than MG that might interfere with the accuracy of study assessments.

Additional, more specific criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Momenta General Queries, Study Director — Momenta Pharmaceuticals, Inc.
Locations (56):
- United States (29):
  - Momenta Investigational Site, Phoenix, Arizona
  - Momenta Investigational Site, Tucson, Arizona
  - Momenta Investigational Site, Los Angeles, California
  - Momenta Investigational Site, Orange, California
  - Momenta Investigational Site, Stanford, California
  - Momenta Investigational Site, Aurora, Colorado
  - Momenta Investigational Site, New Haven, Connecticut
  - Momenta Investigational Site, Boca Raton, Florida
  - Momenta Investigational Site, Maitland, Florida
  - Momenta Investigational Site, Port Charlotte, Florida
  - Momenta Investigational Site, St. Petersburg, Florida
  - Momenta Investigational Site, Augusta, Georgia
  - Momenta Investigational Site, Meridian, Idaho
  - Momenta Investigational Site, Lake Barrington, Illinois
  - Momenta Investigational Site, Fairway, Kansas
  - Momenta Investigational Site, Boston, Massachusetts
  - Momenta Investigational Site, Detroit, Michigan
  - Momenta Investigational Site, East Lansing, Michigan
  - Momenta Investigational Site, Columbia, Missouri
  - Momenta Investigational Site, New Brunswick, New Jersey
  - Momenta Investigational Site, New York, New York
  - Momenta Investigational Site, Charlotte, North Carolina
  - Momenta Investigational Site, Durham, North Carolina
  - Momenta Investigational Site, Raleigh, North Carolina
  - Momenta Investigational Site, Cincinnati, Ohio
  - Momenta Investigational Site, Columbus, Ohio
  - Momenta Investigational Site, Cordova, Tennessee
  - Momenta Investigational Site, Austin, Texas
  - Momenta Investigational Site, Round Rock, Texas
- Belgium (3):
  - Momenta Investigational Site, Leuven, Vlaams Brabant
  - Momenta Investigational Site, Antwerp
  - Momenta Investigational Site, Brussels
- Canada (4):
  - Momenta Investigational Site, Edmonton, Alberta
  - Momenta Investigational Site, London, Ontario
  - Momenta Investigational Site, Toronto, Ontario
  - Momenta Investigational Site, Québec, Quebec
- Germany (4):
  - Momenta Investigational Site, Göttingen, Lower Saxony
  - Momenta Investigational Site, Düsseldorf
  - Momenta Investigational Site, Gummersbach
  - Momenta Investigational Site, Münster
- Italy (3):
  - Momenta Investigational Site, Cefalù
  - Momenta Investigational Site, Messina
  - Momenta Investigational Site, Milan
- Poland (3):
  - Momenta Investigational Site, Krakow
  - Momenta Investigational Site, Lodz
  - Momenta Investigational Site, Warsaw
- Spain (7):
  - Momenta Investigational Site, Barcelona, Catalan
  - Momenta Investigational Site, Badalona, Catalonia
  - Momenta Investigational Site, L'Hospitalet de Llobregat, Catalonia
  - Momenta Investigational Site, Donostia / San Sebastian, Gipuzkoa
  - Momenta Investigational Site, Madrid
  - Momenta Investigational Site, Seville
  - Momenta Investigational Site, Valencia
- United Kingdom (3):
  - Momenta Investigational Site, Birmingham
  - Momenta Investigational Site, Sheffield
  - Momenta Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antozzi C, Guptill J, Bril V, Gamez J, Meuth SG, Nowak RJ, Quan D, Sevilla T, Jouvin MH, Jin J, Karcher K, Ramchandren S, Sun H, Ling L, Zhu Y, Arroyo S; Vivacity-MG Phase 2 Study Group. Safety and Efficacy of Nipocalimab in Patients With Generalized Myasthenia Gravis: Results From the Randomized Phase 2 Vivacity-MG Study. Neurology. 2024 Jan 23;102(2):e207937. doi: 10.1212/WNL.0000000000207937. Epub 2023 Dec 21. PMID 38165333

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received intravenous (IV) infusion of placebo matching to nipocalimab once every 2 weeks (Q2W) starting Day 1 up to Day 57.
- Nipocalimab (M281) 5 Milligrams/Kilogram (mg/kg): Participants received IV infusion of 5 mg/kg nipocalimab once every 4 weeks (Q4W) starting Day 1 up to Day 57. To maintain blinding, participants received matching placebo on Days 15 and 43.
- Nipocalimab 30 mg/kg: Participants received IV infusion of 30 mg/kg nipocalimab once Q4W starting Day 1 up to Day 57. To maintain blinding, participants received matching placebo on Days 15 and 43.
- Nipocalimab 60 mg/kg: Participants received IV infusion of 60 mg/kg nipocalimab single dose on Day 1. To maintain blinding, participants received matching placebo on Days 15, 29, 43 and 57.
- Nipocalimab 60 mg/kg (Q2W): Participants received IV infusion of 60 mg/kg nipocalimab once Q2W starting Day 1 up to Day 57.
Period: Overall Study
Arm/Group | Placebo | Nipocalimab (M281) 5 Milligrams/Kilogram (mg/kg) | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Started | 14 | 14 | 13 | 13 | 14
Completed | 13 | 14 | 12 | 12 | 14
Not Completed | 1 | 0 | 1 | 1 | 0
Not completed — COVID-19 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Nipocalimab 5 Milligrams/Kilogram (mg/kg): Participants received IV infusion of 5 mg/kg nipocalimab once every 4 weeks (Q4W) starting Day 1 up to Day 57. To maintain blinding, participants received matching placebo on Days 15 and 43.
- Total: Total of all reporting groups
Arm/Group | Placebo | Nipocalimab 5 Milligrams/Kilogram (mg/kg) | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W) | Total
Number analyzed (Participants) | 14 | 14 | 13 | 13 | 14 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 9 | 9 | 8 | 43
  >=65 years | 6 | 5 | 4 | 4 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (17.85) | 54.8 (17.64) | 49 (19.54) | 53.1 (15.4) | 59.9 (15.03) | 55 (17.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 9 | 5 | 37
  Male | 6 | 8 | 4 | 4 | 9 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 13 | 14 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
  Other | 2 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 3 | 1 | 0 | 9
  Not Hispanic or Latino | 10 | 13 | 10 | 11 | 14 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 1 | 0 | 0 | 0 | 0 | 1
  CANADA | 2 | 2 | 0 | 0 | 1 | 5
  GERMANY | 1 | 3 | 1 | 0 | 0 | 5
  ITALY | 2 | 2 | 1 | 0 | 0 | 5
  POLAND | 1 | 2 | 1 | 3 | 1 | 8
  SPAIN | 4 | 0 | 6 | 2 | 3 | 15
  UNITED KINGDOM | 0 | 0 | 0 | 3 | 1 | 4
  UNITED STATES | 3 | 5 | 4 | 5 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE are defined as any AE occurring during or after the initiation of the first infusion of study drug.
Time Frame: Up to Day 113
Population: The safety population included all participants who received any amount of nipocalimab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 Milligrams/Kilogram (mg/kg) | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 14 | 14 | 13 | 13 | 14
Participants | 11 | 12 | 9 | 12 | 12

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as any AE occurring during or after the initiation of the first infusion of study drug. An SAE is defined as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: Up to Day 113
Population: The safety population included all participants who received any amount of nipocalimab or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received IV infusion of placebo matching to nipocalimab once Q2W starting Day 1 up to Day 57.
- Nipocalimab 5 mg/kg: Participants received IV infusion of 5 mg/kg nipocalimab once Q4W starting Day 1 up to Day 57. To maintain blinding, participants received matching placebo on Days 15 and 43.
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 14 | 14 | 13 | 13 | 14
Participants | 2 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as any AE occurring during or after the initiation of the first infusion of study drug. For this study, any common terminology criteria for adverse events (CTCAE) Grade 3 or higher event of severe infection or hypoalbuminemia was considered as AESI.
Time Frame: Up to Day 113
Population: The safety population included all participants who received any amount of nipocalimab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 14 | 14 | 13 | 13 | 14
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Change From Baseline to Day 57 in the Myasthenia Gravis - Activities of Daily Living (MG-ADL) Total Score
Description: The MG-ADL was used to assess the participant's MG symptom severity. It assesses eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, and eyelid droop) which were rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score is the sum of the eight function scores and ranges from 0 to 24. Higher scores indicated greater symptom severity/difficulty in performing daily living activities.
Time Frame: Baseline to Day 57
Population: Intent-to-Treat (ITT) population included all randomized participants. Here 'N' (number of participants analyzed) included all participants who were evaluated for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 14 | 12 | 13 | 14
score on a scale | -1.8 (3.22) | -2.5 (2.41) | -3.9 (3.00) | -1.5 (2.82) | -3.9 (3.66)

5. Secondary Outcome: Change From Baseline in Total MG-ADL Score as a Function of Total Serum Immunoglobulin G (IgG) at Day 57
Description: Estimate of additional change from baseline in MG-ADL total score for every 10 percent (%) additional reduction in IgG based on a linear regression of change from baseline in MG-ADL total score on percent reduction in IgG at Day 57. The MG-ADL was used to assess the participant's MG symptom severity. It assesses eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, and eyelid droop) which were rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score is the sum of the eight function scores and ranges from 0 to 24. Higher scores indicated greater symptom severity/difficulty in performing daily living activities.
Time Frame: Baseline and Day 57
Population: All participants over all arms with both an MG-ADL score and an IgG result at both baseline and Day 57 are included in the analysis. Participants are combined over all groups because the analysis correlates MG-ADL change with IgG change and arm was not included as a factor in the pre-specified analysis. Therefore, results by arm are not available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale per 10% IgG reduction
Groups:
- Placebo/Nipocalimab (All Participants): All participants combined over all arms received IV infusion either of placebo or nipocalimab (5 mg/kg [once Q4W]/30 mg/kg[once Q4W]/60 mg/kg[once Q4W]/60 mg/kg [once Q2W]) starting Day 1 up to Day 57.
Arm/Group | Placebo/Nipocalimab (All Participants)
Number analyzed (Participants) | 58
score on a scale per 10% IgG reduction | -0.30 (0.136)

6. Secondary Outcome: Change From Baseline in Total MG-ADL Score as a Response to Percent Change in Total Serum IgG, for Participants Positive for Anti-acetylcholine Receptor (Anti-AChR) Antibodies, at Day 57
Description: Estimate of additional change from baseline in MG-ADL total score for every 10% additional reduction in IgG based on a linear regression of change from baseline in MG-ADL total score on percent reduction in IgG at Day 57 in anti-AChR positive participants. The MG-ADL was used to assess participant's MG symptom severity. It assesses eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, and eyelid droop) which were rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). Total score is sum of eight function scores and ranges from 0 to 24. Higher scores indicated greater symptom severity/difficulty in performing daily living activities.
Time Frame: Baseline and Day 57
Population: All anti-AChR positive participants over all arms with both an MG-ADL score and an IgG result at both baseline and Day 57 are included in the analysis. Participants are combined over all groups because the analysis correlates MG-ADL change with IgG change and arm was not included as a factor in the pre-specified analysis. Therefore, results by arm are not available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale per 10% IgG reduction
Groups:
- Placebo/Nipocalimab (All Anti-AChR Positive Participants): All anti-AChR positive participants combined over all arms received IV infusion of either placebo or nipocalimab (5 mg/kg [once Q4W]/30 mg/kg[once Q4W]/60 mg/kg[once Q4W]/60 mg/kg [once Q2W]) starting Day 1 up to Day 57.
Arm/Group | Placebo/Nipocalimab (All Anti-AChR Positive Participants)
Number analyzed (Participants) | 55
score on a scale per 10% IgG reduction | -0.33 (0.144)

7. Secondary Outcome: Change From Baseline in Total Quantitative Myasthenia Gravis (QMG) Score as a Function of Total Serum IgG at Day 57
Description: Estimate of additional change from baseline in QMG total score for every 10% additional reduction in IgG based on a linear regression of change from baseline in QMG total score on percent reduction in IgG at Day 57. The QMG test was used to assess the participant's strength. The quantitative results of each of the 13 strength components were mapped to a 4-point scale where 0 equals to (=) none, 1= mild, 2= moderate and 3= severe. The total score is the sum of the 13 scale scores and ranges from 0 to 39. Higher scores indicated more severe impairment.
Time Frame: Baseline and Day 57
Population: All participants over all arms with both an QMG score and an IgG result at both baseline and Day 57 are included in the analysis. Participants are combined over all groups because the analysis correlates QMG change with IgG change and arm was not included as a factor in the pre-specified analysis. Therefore, results by arm are not available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale per 10% IgG reduction
Groups:
- Placebo/Nipocalimab (All Participants): All participants combined over all arms received IV infusion of either placebo or nipocalimab (5 mg/kg [once Q4W]/30 mg/kg[once Q4W]/60 mg/kg[once Q4W]/60 mg/kg [once Q2W]) starting Day 1 up to Day 57.
Arm/Group | Placebo/Nipocalimab (All Participants)
Number analyzed (Participants) | 58
score on a scale per 10% IgG reduction | -0.38 (0.174)

8. Secondary Outcome: Change From Baseline in Total QMG Score as a Response to Percent Change in Total Serum IgG, for Participants Positive for Anti-acetylcholine Receptor (Anti-AChR) Antibodies, at Day 57
Description: Estimate of additional change from baseline in QMG total score for every 10% additional reduction in IgG based on a linear regression of change from baseline in QMG total score on percent reduction in IgG at Day 57 in anti-AChR positive participants. The QMG test was used to assess the participant's strength. The quantitative results of each of the 13 strength components were mapped to a 4-point scale where 0 equals to (=) none, 1= mild, 2= moderate and 3= severe. The total score is the sum of the 13 scale scores and ranges from 0 to 39. Higher scores indicated more severe impairment.
Time Frame: Baseline and Day 57
Population: All anti-AChR positive participants over all arms with both an QMG score and an IgG result at both baseline and Day 57 are included in the analysis. Participants are combined over all groups because the analysis correlates QMG change with IgG change and arm was not included as a factor in the pre-specified analysis. Therefore, results by arm are not available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale per 10% IgG reduction
Arm/Group | Placebo/Nipocalimab (All Anti-AChR Positive Participants)
Number analyzed (Participants) | 55
score on a scale per 10% IgG reduction | -0.45 (0.181)

9. Secondary Outcome: Number of Participants With a 2-, 3-, 4-, 5-, 6-, 7-, or Greater Than or Equal to (>=) 8-point Improvement in Total MG-ADL Score at Day 57
Description: as for outcome 4
Time Frame: Day 57
Population: Population analyzed included ITT participants for whom data was available at Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 14 | 12 | 13 | 14
Participants
  2-point Improved | 7 | 9 | 10 | 7 | 12
  3-point Improved | 5 | 9 | 8 | 5 | 11
  4-point Improved | 1 | 5 | 5 | 3 | 7
  5-point Improved | 1 | 2 | 5 | 2 | 6
  6-point Improved | 1 | 1 | 3 | 1 | 3
  7-point Improved | 1 | 1 | 3 | 0 | 2
  >=8-point Improved | 1 | 0 | 1 | 0 | 2

10. Secondary Outcome: Change From Baseline in Total QMG Score at Day 57
Description: The QMG test was used to assess the participant's strength. The quantitative results of each of the 13 strength components were mapped to a 4-point scale where 0 equals to (=) none, 1= mild, 2= moderate and 3= severe. The total score is the sum of the 13 scale scores and ranges from 0 to 39. Higher scores indicated more severe impairment.
Time Frame: Baseline and Day 57
Population: ITT population included all randomized participants. Here 'N' (number of participants analyzed) included all participants who were evaluated for this OM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 13 | 10 | 11 | 13
score on a scale | -3.7 (2.94) | -3.5 (4.10) | -4.1 (3.45) | -1.5 (2.54) | -5.9 (5.30)

11. Secondary Outcome: Number of Participants With a 3-, 4-, 5-, 6-, 7-, or >= 8-point Improvement in Total QMG Score at Day 57
Description: as for outcome 10
Time Frame: Day 57
Population: Population analyzed included ITT participants for whom data was available at Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 13 | 10 | 11 | 13
Participants
  3-point Improved | 8 | 6 | 6 | 4 | 10
  4-point Improved | 5 | 5 | 6 | 3 | 10
  5-point Improved | 5 | 5 | 5 | 1 | 8
  6-point Improved | 2 | 5 | 4 | 1 | 5
  7-point Improved | 2 | 5 | 1 | 0 | 3
  >= 8-point Improved | 2 | 3 | 1 | 0 | 3

12. Secondary Outcome: Change From Baseline in Total Revised Myasthenia Gravis Quality of Life - 15 (MG-QoL-15r) Scale Score at Day 57
Description: The MG-QoL15r was used to assess the participant's limitations related to living with MG. Each of the 15 questions were rated by the participant on a 3-point scale (0= Not at all, 1= somewhat, 2=very much) based on a recall period of "over the past few weeks". The total score is the sum of the 15 question scores and ranges from 0 to 30. Higher scores indicated more limitation.
Time Frame: Baseline and Day 57
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 14 | 12 | 13 | 14
score on a scale | -2.0 (4.58) | -1.7 (4.16) | -6.8 (5.73) | -1.2 (1.91) | -3.7 (5.37)

13. Secondary Outcome: Change From Baseline in Total Serum IgG at Day 57
Description: Change from baseline in total serum IgG was reported. Blood samples were collected for analysis of total serum IgG.
Time Frame: Baseline and Day 57
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: gram/liter (g/L)
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 13 | 10 | 11 | 13
gram/liter (g/L) | -0.3 (1.82) | -1.5 (1.01) | -3.4 (1.01) | -1.7 (1.23) | -7.6 (2.27)

14. Secondary Outcome: Change From Baseline in Total MG-ADL Score at Day 85 and Day 113
Description: as for outcome 4
Time Frame: Baseline, Day 85 and Day 113
Population: ITT population included all randomized participants. Here 'N' (number of participants analyzed) included all participants who were evaluated for this OM and 'n' (number analyzed) included the number of participants evaluated for specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 14
score on a scale
  Day 85: number analyzed (Participants) | 11 | 14 | 11 | 13 | 14
  Day 85 | -2.2 (2.64) | -2.1 (2.40) | -3.7 (2.69) | -1.9 (2.29) | -3.6 (2.79)
  Day 113: number analyzed (Participants) | 12 | 14 | 12 | 12 | 14
  Day 113 | -2.6 (3.09) | -1.0 (2.25) | -2.8 (2.33) | -2.4 (2.78) | -2.6 (3.30)

15. Secondary Outcome: Change From Baseline in Total QMG Score at Day 85 and Day 113
Description: as for outcome 10
Time Frame: Baseline, Day 85 and Day 113
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Nipocalimab 5 Milligram/Kilogram (mg/kg): Participants received IV infusion of 5 mg/kg nipocalimab once Q4W starting Day 1 up to Day 57. To maintain blinding, participants received matching placebo on Days 15 and 43.
Arm/Group | Placebo | Nipocalimab 5 Milligram/Kilogram (mg/kg) | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 14 | 10 | 9 | 13
score on a scale
  Day 85: number analyzed (Participants) | 10 | 13 | 9 | 9 | 13
  Day 85 | -4.0 (2.62) | -3.6 (3.23) | -4.8 (2.49) | -2.0 (2.60) | -5.1 (3.52)
  Day 113: number analyzed (Participants) | 9 | 14 | 10 | 9 | 12
  Day 113 | -4.7 (3.04) | -2.1 (2.40) | -4.2 (3.08) | -3.2 (2.28) | -3.3 (5.69)

16. Secondary Outcome: Change From Baseline in Total MG-QoL15r Score at Day 85 and Day 113
Description: as for outcome 12
Time Frame: Baseline, Day 85 and Day 113
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 13
score on a scale
  Day 85: number analyzed (Participants) | 11 | 14 | 11 | 13 | 13
  Day 85 | -2.5 (2.84) | -2.9 (3.74) | -6.5 (5.66) | -0.7 (4.25) | -3.5 (5.61)
  Day 113: number analyzed (Participants) | 12 | 14 | 12 | 12 | 13
  Day 113 | -3.2 (3.90) | -1.6 (4.20) | -4.2 (4.32) | -1.0 (2.92) | -2.5 (6.09)

17. Secondary Outcome: Number of Participants With Shift From Baseline in Myasthenia Gravis Foundation of America (MGFA) Classification at Day 57
Description: The MGFA was used to assess the participant's MG severity. MGFA classification identifies the subgroup participants with MG who share distinct clinical features or severity of disease: Class I (ocular MG), classes II, III and IV generalized MG with mild, moderate and severe disease, respectively; Class V MG crisis. Separate subclasses under classes II, III and IV are designed: "a" if the predominant weakness is affecting limb/axial weakness or both; subclass "b" if the predominant weakness is affecting oropharyngeal or respiratory muscles or both. In the MGFA classification, lower roman numerals mean less severity. Changes in MGFA classification (regardless of subclass) are categorized as "Improved" (example, III to II), "Same" (example, II to II), or "Worsened" (example, II to III).
Time Frame: Baseline and Day 57
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12
Participants
  Improved | 6 | 3 | 7 | 4 | 7
  Same | 6 | 9 | 3 | 8 | 4
  Worsened | 0 | 0 | 1 | 0 | 1

18. Secondary Outcome: Number of Participants With Shift From Baseline in MGFA Classification to Day 113
Description: as for outcome 17
Time Frame: Baseline to Day 113
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 11
Participants
  Improved | 3 | 2 | 3 | 2 | 3
  Same | 6 | 5 | 4 | 5 | 5
  Worsened | 0 | 2 | 1 | 0 | 3

19. Secondary Outcome: Change From Baseline in Total Serum IgG at Day 85 and Day 113
Description: Change from baseline in total serum IgG at Day 85 and Day 113 was analyzed. Blood samples were collected for analysis of total serum IgG.
Time Frame: Baseline, Day 85 and Day 113
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 14 | 11 | 9 | 13
g/L
  Day 85: number analyzed (Participants) | 11 | 13 | 10 | 9 | 13
  Day 85 | -0.5 (1.02) | -1.4 (1.93) | -3.8 (1.28) | -1.2 (1.02) | -5.7 (2.30)
  Day 113: number analyzed (Participants) | 10 | 14 | 11 | 9 | 12
  Day 113 | -0.6 (1.19) | -0.7 (1.48) | -1.2 (0.78) | -0.7 (1.09) | -2.2 (1.73)

20. Secondary Outcome: Serum Concentrations of Nipocalimab
Description: Serum concentrations of nipocalimab were reported. Concentrations below the lowest quantifiable concentration (< LLOQ) that is <0.15 microgram/milliliter (mcg/mL) was treated as zero in calculating the summary statistics.
Time Frame: Baseline (Pre Infusion and Post Infusion), Day 15 (Pre Infusion), Day 29 (Pre Infusion), Day 43 (Pre Infusion), Day 57 (Pre Infusion and Post Infusion) and Day 85
Population: The safety population included all participants who received any amount of nipocalimab or placebo. Here 'n' (number analyzed) included the number of participants evaluated for specific timepoints.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Nipocalimab 5 mg/kg | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
Number analyzed (Participants) | 14 | 13 | 13 | 14
micrograms/milliliter (mcg/mL)
  Baseline (Pre Infusion) | 0.0 (0.005) | 0.00 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Baseline (Post Infusion): number analyzed (Participants) | 4 | 5 | 4 | 5
  Baseline (Post Infusion) | 117.75 (84.835) | 746.80 (47.214) | 1847.50 (153.270) | 1325.00 (616.443)
  Day 15 (Pre Infusion) | 0.0 (0.006) | 0.01 (0.010) | 27.61 (42.167) | 29.30 (36.631)
  Day 29 (Pre Infusion): number analyzed (Participants) | 14 | 10 | 11 | 14
  Day 29 (Pre Infusion) | 0.0 (0.004) | 0.0 (0.0) | 0.0 (0.0) | 72.69 (152.058)
  Day 43 (Pre Infusion): number analyzed (Participants) | 14 | 12 | 11 | 14
  Day 43 (Pre Infusion) | 0.0 (0.004) | 0.01 (0.013) | 0.0 (0.0) | 66.72 (85.919)
  Day 57 (Pre Infusion): number analyzed (Participants) | 13 | 10 | 11 | 13
  Day 57 (Pre Infusion) | 0.0 (0.006) | 95.40 (301.681) | 0.0 (0.0) | 44.80 (68.560)
  Day 57 (Post Infusion): number analyzed (Participants) | 2 | 2 | 3 | 4
  Day 57 (Post Infusion) | 49.15 (41.507) | 746.50 (96.874) | 0.0 (0.0) | 1827.50 (741.052)
  Day 85: number analyzed (Participants) | 13 | 10 | 9 | 13
  Day 85 | 0.0 (0.007) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.004)

ADVERSE EVENTS:
Time Frame: Up to Day 113
Description: The safety population included all participants who received any amount of nipocalimab or placebo.
Arm/Group | Placebo | Nipocalimab 5 Milligrams/Kilogram (mg/kg) | Nipocalimab 30 mg/kg | Nipocalimab 60 mg/kg | Nipocalimab 60 mg/kg (Q2W)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/14 | 1/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 10/14 | 12/14 | 8/13 | 12/13 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Nipocalimab 5 Milligrams/Kilogram (mg/kg) (N=14) | Nipocalimab 30 mg/kg (N=13) | Nipocalimab 60 mg/kg (N=13) | Nipocalimab 60 mg/kg (Q2W) (N=14)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myasthenia Gravis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Nipocalimab 5 Milligrams/Kilogram (mg/kg) (N=14) | Nipocalimab 30 mg/kg (N=13) | Nipocalimab 60 mg/kg (N=13) | Nipocalimab 60 mg/kg (Q2W) (N=14)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid Ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Feeling Cold (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 1 | 2
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Vessel Puncture Site Pruritus (General disorders) | 0 | 0 | 0 | 0 | 1
Vessel Puncture Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Asymptomatic Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Palate Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Bacterial Test (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 1
Carbohydrate Antigen 19-9 Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Helicobacter Test Positive (Investigations) | 1 | 0 | 0 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Neutrophil Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil Percentage Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urine Analysis Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Mononeuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myasthenia Gravis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Brachiocephalic Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Limitations to this study include the small sample sizes of each treatment arm and the study activity disruption due to the COVID-19 pandemic, especially the missed Quantitative Myasthenia Gravis (QMG) assessments which hampered the analysis of the endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03772587/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03772587/SAP_001.pdf